CLINICAL TRIAL: NCT05624281
Title: Expanded Access Program of OFEV® (Nintedanib) in Children and Adolescents (6- to 17-year-old) With Clinically Significant Fibrosing Interstitial Lung Disease (ILD)
Brief Title: A Treatment Protocol to Support the Care of Children and Adolescents With Fibrosing Interstitial Lung Disease (ILD)
Status: No longer available | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0511
Record Dates: First submitted 2022-11-04; First posted 2022-11-22 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lung Diseases, Interstitial (in Pediatric Populations); Childhood Interstitial Lung Disease (chILD)
MeSH Terms: conditions — Lung Diseases | interventions — nintedanib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: nintedanib — nintedanib, for patients with fibrosing interstitial lung disease (ILD); in this EAP limited to children and adolescents
  Other Names: OFEV®

SUMMARY:
This Expanded Access Program (EAP) is intended to facilitate the availability of OFEV® (nintedanib) to children and adolescents with chronic fibrosing interstitial lung disease (ILD) on top of current standard of care treatment and for whom no satisfactory authorized alternative therapy exists and who cannot participate in the ongoing 1199-0378 trial.

ELIGIBILITY:
Inclusion criteria:

* Patients who are not eligible or unable to participate in the ongoing 1199-0378 trial.
* Children and adolescents 6 to 17 years old at Visit 1.
* Signed and dated written informed consent and assent, where applicable, in accordance with International Council on Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients. Females of childbearing potential (WOCBP) must confirm that sexual abstinence is standard practice and will be continued until 3 months after last drug intake, or be ready and able to use a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly, in combination with one barrier method, from 28 days prior to initiation of study treatment, during treatment and until 3 months after last drug intake. Sexual abstinence is defined as abstinence from any sexual act that may result in pregnancy. A list of contraception methods meeting these criteria is provided in the parental information and in the protocol.
* Patients with evidence of fibrosing Interstitial Lung Disease (ILD) on high-resolution computed tomography (HRCT) within 12 months of Visit 1 as assessed and documented by the investigator.

Further inclusion criteria for the determination of fibrosing ILD on HRCT are defined in the protocol.

* Patients with Forced Vital Capacity (FVC) % predicted ≥25% at Visit 1.
* Patients with clinically significant disease at Visit 1, as assessed by the investigator:

  * Fan score >3
  * Documented evidence of clinical progression over time based on either

    * a 5-10% relative decline in FVC% predicted accompanied by worsening symptoms, or
    * a ≥10% relative decline in FVC % predicted, or
    * increased fibrosis on HRCT, or
    * other measures of clinical worsening attributed to progressive lung disease (e.g., increased oxygen requirement, decreased diffusion capacity).

Exclusion criteria

* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the program.
* Currently enrolled in another investigational device or drug program, or less than 30 days since ending another investigational device or drug program(s) or receiving other investigational treatment(s). This does not apply to nintedanib.
* Women who are pregnant, nursing, or who plan to become pregnant while in the program.
* Aspartate Transaminase (AST) and/or Alanine Aminotransferase (ALT) >1.5 x Upper Level of Normal (ULN) at Visit 1.
* Bilirubin >1.5 x ULN at Visit 1.
* Estimated Glomerular Filtration Rate (eGFR) <30 mL/min calculated by Schwartz formula at Visit 1.
* Patients with underlying chronic liver disease (Child Pugh A, B or C hepatic impairment) at Visit 1.
* Other investigational therapy received within 1 month or 5 half-lives (whichever is greater but ≥1 week) prior to Visit 1.

Further exclusion criteria apply.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com